CLINICAL TRIAL: NCT03762902
Title: The Relation Between Analyzed Sensory Data of the Smartphone and Migraine Attacks, Recorded by Individuals Who Suffer From Episodic Migraine
Brief Title: Predicting Migraine Attacks Based on Environmental and Behavioral Changes as Detected From the Smartphone
Acronym: Migraine
Status: Terminated | Type: Observational
Why Stopped: Sufficient data was collected through the app to achieve initial results
Sponsor: Lifegraph Ltd. (Industry)
Collaborators: Henry Ford Health System (Other)
Responsible Party: Sponsor
Other Study IDs: LifegraphMigrainePrediction
Record Dates: First submitted 2018-11-30; First posted 2018-12-04 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-05

CONDITIONS: Migraine Disorders; Headache Disorders; Headache Disorders, Primary; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases
Keywords: Migraine; Smartphone; App; Prediction; Forecast; Detection; Individual; Machine Learning; Data Science; Algorithm; Behavior; Henry Ford Health System; HFHS; Lifegraph
MeSH Terms: conditions — Migraine Disorders; Headache Disorders; Headache Disorders, Primary; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Alzheimer Disease; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is conducted at the Henry Ford Health System with Lifegraph's behavioral monitoring technology, to examine the relation between migraine attacks and behavioral and environmental changes as detected from the smartphone sensors. The investigators hypothesize that Lifegraph's technology can predict the occurrence of migraine attacks with high precision.

DETAILED DESCRIPTION:
Migraine attacks can damage quality of life and lead to missed work days if not treated in time. These attacks last for about 4-72 hours, accompanied by headache and other symptoms. The time window for early intervention, which can potentially reduce the severity of an attack, lasts 2-48 hours before symptoms are starting to appear (10 hours on average). This time window is defined in the literature as the prodromal phase, when intervention during this phase can allow early treatment to improve the patient's condition and reduce the intensity and duration of the attack.

Migraine attacks and the prodromal phase can be characterized by one or more behavioral or environmental symptoms, either causal or resultant. Some of them can be passively measured by the smartphone usage, such as changes in sleep, physical activity and weather.

Lifegraph's smartphone application runs in the background of the subjects' personal smartphone, collects data passively and automatically, while rigorously maintaining privacy and with no effect to the daily use. Proprietary machine-learning algorithms analyze the collected data and turn it into behavioral channels, such as activity, sleep and mobility. The technology learns the personal routine of each user and detects changes in his/her behavioral patterns that can indicate an upcoming migraine.

Eligible subjects will meet a neurologist, sign an informed consent, fill an initial questionnaire and install the Lifegraph application on their smartphone. The application requires a one-time registration process.

During the study, subjects will self-report migraine attacks they experience through the smartphone application. Each report will include start time, end time and pain intensity. Data will be analyzed during the study in order to learn each subject's behavior and his/her migraine attacks. Subjects will be blinded to the app's migraine predictions to avoid expectancy bias.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who suffer from episodic migraine with 4-14 days of migraine per month (ICHD-3 patients).
* Individuals who possess a smartphone - Android version 5.0 and above or iOS version 10.0 and above.

Exclusion Criteria:

* Individuals who are unable to sign the consent form.
* Pregnant women.
* Individuals suffering from headaches that do not meet the IHS migraine criteria or don't have moderate to severe chronic pain of VAS chronic grade 4 and above.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who suffer from episodic migraine
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Assessing Lifegraph's predictive ability of migraine attacks before subjects report they experience an attack. | 3 months
  Lifegraph has created a scalable and dynamic platform to accommodate different conditions, different types of patients with different types of data, concurrently. This platform converts the raw sensor data accumulating in Lifegraph's servers into behavioral and environmental features that have been found to be informative and helpful in generating insights relevant to migraines. The features are fed into machine learning algorithms that search for early signs of change, that may indicate an oncoming attack. These algorithms may be divided into population-based and personalized models. The study will develop a separate predictive model for each subject to predict the probability of experiencing a migraine attack during a particular interval (e.g. the next 12, 24, or 48 hours). Higher precision values of prediction will represent a better outcome. The precision is expected to be 50-70%, depends on the time passed since first installing the app and the number of reported migraine attacks

CONTACTS AND LOCATIONS:
Overall Officials: Ashhar Ali, DO, Principal Investigator — Senior Staff Physician, Department of Neurology
Locations (2):
- United States (2):
  - Henry Ford Health System Main Campus, Detroit, Michigan
  - Henry Ford Health System, West Bloomfield, Michigan

IPD SHARING:
Plan to Share IPD: No